CLINICAL TRIAL: NCT01696461
Title: A Phase II Study Evaluating the Safety and Efficacy of Subcutaneous Plerixafor for the Mobilization and Transplantation of HLA-Matched Sibling Donor Hematopoietic Stem Cells in Recipients With Hematological Malignancies
Brief Title: A Phase II Study Evaluating the Safety and Efficacy of Subcutaneous Plerixafor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: Genzyme, a Sanofi Company (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-PLEX
Record Dates: First submitted 2012-09-24; First posted 2012-10-01 (Estimated); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-05

CONDITIONS: Related Donors Donating Peripheral Blood Stem Cells (PBSC) to a Family Member; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Chronic Myelogenous Leukemia; Non-Hodgkin's Lymphoma; Hodgkin's Disease; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Related donors receiving plerixafor (Experimental): Collection of sufficient CD34+ cells using plerixafor as the mobilizing agent.
  Eligible donors determined according to institutional standards
  * 18-65 years of age
  * 6/6 HLA-matched sibling
  * Fulfill individual Transplant Center criteria to serve as a mobilized blood cell donor
  * Serum creatinine <1.5 x institution upper limit of normal (ULN) or estimated creatinine clearance (CLCR) >50 mL/min
  Treatment Description:
  * Receive subcutaneous plerixafor at 240 μg/kg and commence leukapheresis approximately 4 hours later.
  * Leukapheresis will be performed up to two consecutive days. The target CD34+ cell dose is > 4.0 x 106/kg with a minimum of > 2.0 x 106/kg.
  Interventions: Drug: Plerixafor
- Recipients, myeloablative regimen (No Intervention): Patients undergoing conditioning under a myeloablative regimen
  Myeloablative (one of four general regimens):
  Busulfan (> 9 mg/kg po or iv total) with fludarabine Busulfan (> 9 mg/kg po or iv total) with cyclophosphamide Total body irradiation (> 1000 cGy) plus etoposide Total body irradiation (> 500 cGy) plus cyclophosphamide
- Recipients, reduced intensity conditioning regimen. (No Intervention): Patients undergoing conditioning using a reduced intensity conditioning regimen.
  Reduced Intensity (one of three general regimens):
  Busulfan (< 9 mg/kg po or iv total) plus fludarabine Melphalan (100-140 mg/m2 iv total) plus fludarabine Fludarabine plus cyclophosphamide (> 2000 mg/m2 total)

INTERVENTIONS:
Drug: Plerixafor
  Other Names: Mozobil; AMD3000
  Arms: Related donors receiving plerixafor

SUMMARY:
This is a Phase II, open-label, two strata, multicenter, prospective study of plerixafor-mobilized HLA-identical sibling allografts in recipients with hematological malignancies. This study will establish the safety and efficacy of subcutaneous plerixafor for this purpose.

DETAILED DESCRIPTION:
The primary objective is to determine the proportion of donors whose cells can be successfully mobilized and collected with a sufficient CD34+ cell dose using plerixafor as the mobilizing agent, using an intention-to-treat analysis. Donor mobilization following plerixafor will be considered successful if ≥ 2.0x10e6 CD34+ cells/kg recipient weight are collected in no more than two leukapheresis collections.

All donors receiving plerixafor will be included in the analysis of the primary objective based on the intention-to-treat principle.Recipients will be classified into one of the two strata, myeloablative or reduced intensity, according to his/her conditioning regimen. The target enrollment is 64 donor/recipient pairs, 32 pairs per stratum.

ELIGIBILITY:
Inclusion Criteria:

Donor:

* Donor eligibility will be determined according to applicable federal, state and local regulations and institutional standards
* 18-65 years of age
* 6/6 HLA-matched sibling
* Fulfill individual Transplant Center criteria to serve as a mobilized blood cell donor
* Serum creatinine <2.0mg/dl

Recipient:

* 18 to 65 years of age
* 6/6 HLA antigen matched sibling willing to donate PBSC for transplant
* Fulfill individual Transplant Center Criteria for transplant
* One of the following diagnoses:

  * Acute myelogenous leukemia (AML) in 1st remission or beyond with <5% marrow blasts and no circulating blasts. Marrow must be done within 30 days of the start of transplant conditioning regimen in alignment with other pre-transplant assessments.
  * Acute lymphoblastic leukemia (ALL) in 1st remission or beyond with <5% marrow blasts and no circulating blasts
  * Myelodysplastic syndrome, either intermediate-1,2, or high risk by International Prognostic Scoring System or transfusion dependent
  * Chronic myelogenous leukemia (CML) failing or intolerant to tyrosine kinase inhibitor based therapy
  * Non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD) in 2nd or greater complete remission, partial remission, or in relapse (but with at least stable disease after most recent therapy)
  * Chronic lymphocytic leukemia (CLL), relapsing after at least one prior regimen, or in remission with 17p deletion
* Serum creatinine must be <2.0mg/dl
* Total bilirubin and aspartate aminotransferase (AST) <3x normal
* Infectious disease marker (IDM) monitoring will be performed per institutional standards
* Karnofsky performance status of 70% or greater.
* Patients who have undergone a prior autologous transplantation are eligible for a reduced intensity transplant only

Exclusion Criteria:

Donor:

* Donor unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
* Donor already enrolled on another investigational agent study
* Pregnant or breast feeding females, or females not willing or able to use adequate contraception if sexually active

Recipient:

* Patient unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
* Patients with active, uncontrolled infection at the time of the transplant preparative regimen
* Pregnant or breast feeding females, or females not willing or able to use adequate contraception if sexually active
* Patients with a history of previous central nervous system (CNS) tumor involvement showing active symptoms or signs along with documented disease on lumbar puncture and MRI of the brain within 30 days of start of conditioning
* A condition, which, in the opinion of the clinical investigator, would interfere with the evaluation of primary and secondary endpoints.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2013-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Devine, MD, Principal Investigator — NMDP/BeTheMatch
Locations (12):
- United States (12):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Chen YB, Le-Rademacher J, Brazauskas R, Kiefer DM, Hamadani M, DiPersio JF, Litzow MR, Craig M, Horwitz ME, Artz AS, McClune BL, Fernandez HF, Duong HK, Kobusingye H, Proue M, Drexler RJ, Horowitz MM, Shaw BE, Miller JP, Hosoba S, Waller EK, Devine SM. Plerixafor alone for the mobilization and transplantation of HLA-matched sibling donor hematopoietic stem cells. Blood Adv. 2019 Mar 26;3(6):875-883. doi: 10.1182/bloodadvances.2018027599. PMID 30890544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible donor-recipient pairs were recruited at 12 US hematopoietic cell transplantation (HCT) transplant centers between July 2013 and December 2014. Recipients who met eligibility criteria provided written informed consent prior to any study procedure being performed. In order for the recipient to proceed in the study, intended donors were required to consent as well.
Groups:
- Related Donors Receiving Plerixafor: Collection of sufficient CD34+ cells using plerixafor as the mobilizing agent.
  Donor eligibility was determined according to institutional standards Donors met the following criteria:
  * 18-65 years of age
  * 6/6 HLA-matched sibling
  * Fulfill individual Transplant Center criteria to serve as a mobilized blood cell donor
  * Serum creatinine <1.5 x institution ULN or estimated creatinine clearance (CLCR) >50 mL/min
  Treatment Description:
  * Receive subcutaneous plerixafor at 240 μg/kg and commence leukapheresis approximately 4 hours later.
  * Leukapheresis will be performed up to two consecutive days. The target CD34+ cell dose is > 4.0 x 106/kg with a minimum of > 2.0 x 106/kg.
- Recipients, Reduced Intensity: Reduced Intensity (one of three general regimens):
  Busulfan (< 9 mg/kg po or iv total) plus fludarabine Melphalan (100-140 mg/m2 iv total) plus fludarabine Fludarabine plus cyclophosphamide (> 2000 mg/m2 total).
- Recipients Myeloablative Regimen: Myeloablative (one of four general regimens):
  Busulfan (> 9 mg/kg po or iv total) with fludarabine Busulfan (> 9 mg/kg po or iv total) with cyclophosphamide Total body irradiation (> 1000 cGy) plus etoposide Total body irradiation (> 500 cGy) plus cyclophosphamide
Period: Overall Study
Arm/Group | Related Donors Receiving Plerixafor | Recipients, Reduced Intensity | Recipients Myeloablative Regimen
Started | 64 (First donor-recipient pair was enrolled in July, 2013.) | 33 | 30
Completed | 64 (Last donor-recipient pair was enrolled in December, 2014) | 33 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Related Donors Receiving Plerixafor: Collection of sufficient CD34+ cells using plerixafor as the mobilizing agent.
  Eligible donors determined according to institutional standards
  * 18-65 years of age
  * 6/6 HLA-matched sibling
  * Fulfill individual Transplant Center criteria to serve as a mobilized blood cell donor
  * Serum creatinine <1.5 x institution ULN or estimated creatinine clearance (CLCR) >50 mL/min
  Treatment Description:
  * Receive subcutaneous plerixafor at 240 μg/kg and commence leukapheresis approximately 4 hours later.
  * Leukapheresis will be performed up to two consecutive days. The target CD34+ cell dose is > 4.0 x 106/kg with a minimum of > 2.0 x 10E6/kg.
- Recipients, Myeloablative Conditioning Regimen: Myeloablative (one of four general regimens):
  Busulfan (> 9 mg/kg po or iv total) with fludarabine Busulfan (> 9 mg/kg po or iv total) with cyclophosphamide Total body irradiation (> 1000 cGy) plus etoposide Total body irradiation (> 500 cGy) plus cyclophosphamide
- Recipients, Reduced Intensity Conditioning Regimen: Reduced Intensity (one of three general regimens):
  Busulfan (< 9 mg/kg po or iv total) plus fludarabine Melphalan (100-140 mg/m2 iv total) plus fludarabine Fludarabine plus cyclophosphamide (> 2000 mg/m2 total)
- Total: Total of all reporting groups
Arm/Group | Related Donors Receiving Plerixafor | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen | Total
Number analyzed (Participants) | 64 | 30 | 33 | 127
Age, Categorical [Count of Participants; unit: Participants] — Donor age at collection, years
  Participants
    <=18 years | 1 | 0 | 0 | 1
    Between 18 and 65 years | 61 | 30 | 30 | 121
    >=65 years | 2 | 0 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Information collected by subject response to questions on case report forms
  Participants
    Female | 23 | 14 | 24 | 61
    Male | 41 | 16 | 9 | 66
Region of Enrollment [Number; unit: participants]
  United States | 64 | 30 | 33 | 127

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Donors Whose Cells Were Successfully Mobilized and Collected With a Sufficient CD34+ Cell Dose Using Plerixafor as the Mobilizing Agent, Using an Intention-to-treat Analysis.
Description: Donor mobilization following plerixafor was considered successful if ≥ 2.0x106 CD34+ cells/kg recipient weight was collected in no more than two leukapheresis collections.
Time Frame: donation
Population: Recipients were not mobilized with plerixafor.
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donors Receiving Plerixafor
Number analyzed (Participants) | 64
Participants | 63
Statistical Analysis 1: Comparison: Related Donors Receiving Plerixafor; Test type: Other; Percentage of donors mobilized with plerixafor. No comparison group was analyzed

2. Secondary Outcome: Incidence and Severity of Acute Toxicities
Description: Incidence and severity of acute toxicities before and during apheresis experienced by donors receiving plerixafor. Acute toxicities are graded according to the NCI Common Terminology Criteria for Adverse Events, version 4.0. This outcome measure is descriptive. Grade of maximum toxicity across all time points is reported. Higher grades denote worse outcomes. 0 = None, 1 = Mild, 2 = Moderate, 3 = severe.
Time Frame: baseline, Day 1, Day 2, Day 3
Population: Recipients were not analyzed for this outcome measure
Measure: Count of Participants; unit: Participants
Groups:
- Related Donors Receiving Plerixafor: Collection of sufficient CD34+ cells using plerixafor as the mobilizing agent.
  Eligible donors determined according to institutional standards
  * 18-65 years of age
  * 6/6 HLA-matched sibling
  * Fulfill individual Transplant Center criteria to serve as a mobilized blood cell donor
  * Serum creatinine <1.5 x institution ULN or estimated creatinine clearance (CLCR) >50 mL/min
  Treatment Description:
  * Receive subcutaneous plerixafor at 240 μg/kg and commence leukapheresis approximately 4 hours later.
  * Leukapheresis will be performed up to two consecutive days. The target CD34+ cell dose is > 4.0 x 106/kg with a minimum of > 2.0 x 106/kg.
  Plerixafor
Arm/Group | Related Donors Receiving Plerixafor
Number analyzed (Participants) | 64
Participants
  Max Modified toxicity criteria (MTC) = 0 | 19
  Max Modified toxicity criteria (MTC) = 1 | 34
  Max Modified toxicity criteria (MTC) = 2 | 10
  Max Modified toxicity criteria (MTC) = 3 | 1
Statistical Analysis 1: Comparison: Related Donors Receiving Plerixafor; Test type: Other; This is a descriptive analysis. Percentage of donor experiencing toxicities was assessed at 30, 60, 120, and 240 minutes after administration of plerixafor on each day of collection and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.3. Grade of maximum toxicity across all time points is reported

3. Secondary Outcome: Adverse Effects
Description: Adverse effects experienced by donors receiving plerixafor up to one year post donation. Number of participants with a maximum MTC >0 reported at each individual time point. Adverse effects are graded according to the NCI Common Terminology Criteria for Adverse Events, version 4.0. This outcome measure is descriptive. Participants can experience adverse effects at more than one time point evaluated. Higher grades denote worse outcomes. 0 = None, 1 = Mild, 2 = Moderate, 3 = severe.
Time Frame: 30 minutes, 60 minutes, 120 minutes, 240 minutes, 1 month, 6 months, 12 months post donation for each subject
Population: Recipients did not receive plerixafor and were not examined for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Related Donors Receiving Plerixafor
Number analyzed (Participants) | 64
Participants
  30 minutes after administration of plerixafor | 23
  60 minutes after administration of plerixafor | 28
  120 minutes after administration of plerixafor | 27
  240 minutes after administration of plerixafor | 24
  One month after administration of plerixafor | 22
  Six months after administration of plerixafor | 7
  Twelve months after administration of plerixafor | 7
Statistical Analysis 1: Comparison: Related Donors Receiving Plerixafor; Test type: Other; This is a descriptive analysis. The number of donors experiencing toxicities was assessed at 30, 60, 120, and 240 minutes after administration of plerixafor on each day of collection and one, six, and 12 months post-donation. Toxicities were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.3

4. Secondary Outcome: Incidence of and Kinetics of Neutrophil and Platelet Recovery After Transplantation of Hematopoietic Cells Mobilized With Plerixafor
Description: Incidence of and kinetics of neutrophil and platelet recovery by day 100 in recipients after transplantation of hematopoietic cells mobilized with plerixafor.
Time Frame: Day +1 through neutrophil recovery or Day 21 (whichever is first)
Population: Patients were classified to one of the two conditioning regimens - myeloablative (MAC) or reduced intensity conditioning (RIC). A total of 30 MAC and 33 RIC patients were analyzed for this outcome. Neutrophil engraftment was defined as time from day 0 of HCT to the first of 3 consecutive measurements of absolute neutrophil count ≥0.5 × 109/L. Platelet engraftment was defined as the number of days from day 0 of HCT to the first of 3 consecutive values of platelet count ≥20 × 109/L.
Measure: Number (95% Confidence Interval); unit: Percentage probability of engraftment
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
Percentage probability of engraftment
  Neutrophil engraftment | 100 [100 to 100] | 100 [100 to 100]
  Platelet engraftment | 100 [100 to 100] | 97 [97 to 100]
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; Test type: Other; At 100 days after HCT, all patients in both the MAC and the RIC cohorts had achieved neutrophil engraftment. All patients in the MAC arm and 97% of patients in the RIC arm had achieved platelet engraftment. The median time to neutrophil engraftment was 13 and 15 days for MAC and RIC, respectively. The median time to platelet engraftment was 19 and 18 days for MAC and RIC, respectively

5. Secondary Outcome: T-cell (CD3+) and Myeloid (CD33+) Chimerism After Transplantation of Hematopoietic Cells Mobilized With Plerixafor
Description: T-cell (CD3+) and myeloid (CD33+) chimerism in recipients after transplantation of hematopoietic cells mobilized with plerixafor. This outcome measure is descriptive.
Time Frame: Chimerism was evaluated at serial timepoints post HCT in patients in both RIC and MAC strata. Chimerism was assessed at Day +28, +100, +180, and +365
Population: Chimerism is not evaluated in donor arm.
Measure: Median (Full Range); unit: percentage of donor cell chimerism
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
percentage of donor cell chimerism
  Myeloid chimerism (Day 28) | 100 [98 to 100] | 100 [91 to 100]
  T-cell chimerism (Day 28) | 92 [59 to 100] | 80 [50 to 100]
  Myeloid chimerism (Day 100) | 99 [91 to 100] | 100 [17 to 100]
  T-cell chimerism (Day 100) | 97 [76 to 100] | 84 [64 to 100]
  Myeloid chimerism (Day 180) | 100 [89 to 100] | 100 [5 to 100]
  T-cell chimerism (Day 180) | 100 [91 to 100] | 95 [5 to 100]
  Myeloid chimerism (Day 365) | 100 [100 to 100] | 100 [0 to 100]
  T-cell chimerism (Day 365) | 100 [100 to 100] | 100 [0 to 100]
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; Test type: Other; Full donor myeloid chimerism was achieved relatively quickly in both RIC and MAC groups (median 100% at day +28 in both RIC and MAC), but conversion to full donor T-cell chimerism appeared to be slower in the RIC patients. T-cell chimerism for MAC patients: median donor cell % (range): Day +28: 92(59-100)%, Day +100: 97(76-100)%, Day +180: 100(91-100)%, Day +365: 100(100-100)% T-cell chimerism for RIC patients: median donor cell % (range): Day +28: 80(50-100)%, Day +100: 84(64-100)%, Day +180: 95(74-100)%, Day +365: 100(87-100)%

6. Secondary Outcome: Primary Graft Failure After Transplantation of Hematopoietic Cells Mobilized With Plerixafor
Description: Incidence of primary graft failure in recipients after transplantation of hematopoietic cells mobilized with plerixafor. This outcome measure is descriptive.
Time Frame: Day 28
Population: Donor population did not receive a transplant
Measure: Count of Participants; unit: Participants
Groups:
- Recipients, Reduced Intensity Conditioning Regimen: Busulfan (< 9 mg/kg po or iv total) plus fludarabine Melphalan (100-140 mg/m2 iv total) plus fludarabine Fludarabine plus cyclophosphamide (> 2000 mg/m2 total)
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
Participants | 0 | 0
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; Test type: Other; This is a descriptive outcome.There were no cases of primary graft failure

7. Secondary Outcome: Incidence of Acute Graft-versus-host Disease (GVHD)
Description: Incidence of acute graft-versus-host disease (GVHD) in recipients after transplantation of hematopoietic cells mobilized with plerixafor
Time Frame: Day 100
Population: Donor arm did not receive a transplant. This group was not analyzed for graft-vs-host disease
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
Percentage of participants
  Grade 2-4 aGVHD by day 100 | 53 [35 to 71] | 18 [7 to 33]
  Grade 3-4 aGVHD by day 100 | 17 [6 to 32] | 3 [0 to 12]
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; The cumulative incidence of acute graft-vs-host disease was examined in the RIC and MAC groups but was not directly compared with a statistical test; Test type: Other; The incidence of acute GVHD was quantified by computing the cumulative incidence probability and an appropriate 95% confidence interval. Death was treated as a competing risk

8. Secondary Outcome: Immune Reconstitution
Description: Rate and quality of immune reconstitution as evidenced by peripheral blood immunophenotype after transplantation of hematopoietic cells mobilized with plerixafor.
Time Frame: Day 28, 100, 180, 365
Population: Donor population did not receive a transplant. Immune reconstitution was not measured in the donor population.
Measure: Median (Full Range); unit: Cells*10^3/mm^3
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
Cells*10^3/mm^3
  CD3+ (Day 28) | 589 [48 to 2250] | 478 [49 to 1485]
  CD4+ (Day 28) | 363 [23 to 1364] | 214 [28 to 676]
  CD8+ (Day 28) | 197 [19 to 837] | 127 [8 to 918]
  CD3+ (Day100) | 647 [61 to 1671] | 529 [40 to 1387]
  CD4+ (Day 100) | 339 [20 to 714] | 265 [25 to 650]
  CD8+ (Day 100) | 242 [12 to 1069] | 162 [13 to 998]
  CD3+ (Day 180) | 638 [58 to 1964] | 699 [69 to 1517]
  CD4+ (Day 180) | 352 [16 to 851] | 257 [18 to 769]
  CD8+ (Day 180) | 272 [26 to 1080] | 219 [37 to 862]
  CD3+ (Day 365) | 794 [62 to 1780] | 1094 [207 to 2448]
  CD4+ (Day 365) | 495 [27 to 932] | 457 [92 to 775]
  CD8+ (Day 365) | 264 [25 to 963] | 460 [106 to 1608]
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; Test type: Other; Immune reconstitution was measured by CD3+CD4+ and CD3+CD8+ T cells in the peripheral blood of patients at days 28, 100, 180, and 365 after HCT. Notably, median CD3+CD4+ cell counts were >200/µL at all times analyzed, including day 28 in both MAC and RIC groups

9. Secondary Outcome: Incidence of Cytomegalovirus (CMV) Reactivation After Transplantation With Cells Mobilized With Plerixafor.
Description: Percentage of recipients with prior CMV infection whose CMV was reactivated after transplantation with cell mobilized with plerixafor
Time Frame: day 365
Population: Donor population did not receive a transplant. Only those with prior infection were eligible to be analyzed for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 15 | 26
Participants | 3 | 6
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; Groups were not directly compared using a statistical test; Test type: Other; Percentage of recipients at-risk for CMV reactivation who experienced a reactivation

10. Secondary Outcome: Treatment-related Mortality and Disease Relapse/Progression
Description: Incidence of treatment-related mortality and disease relapse/progression in recipients after transplantation of hematopoietic cells mobilized with plerixafor
Time Frame: Day 180, 365
Population: Related donors did not receive a transplant and were not examined for this outcome.
Measure: Number (95% Confidence Interval); unit: Percentage probability of outcome
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
Percentage probability of outcome
  Treatment-related mortality (180 days) | 7 [1 to 18] | 3 [0 to 12]
  Treatment-related mortality (365 days) | 17 [6 to 32] | 6 [1 to 17]
  Relapse/progression of disease (180 days) | 30 [15 to 47] | 28 [14 to 45]
  Relapse/progression of disease (365 days) | 30 [15 to 48] | 30 [16 to 47]
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; The probability of treatment-related mortality and disease relapse/progression were examined in the RIC and MAC cohorts but were not directly compared between the two groups using a statistical test; Test type: Other; The incidence of treatment-related mortality and relapse was quantified by computing the cumulative incidence probability and an appropriate 95% confidence interval. When computing the cumulative incidence probability of treatment-related mortality and relapse, relapse and treatment-related mortality, respectively, were considered as a competing risk

11. Secondary Outcome: Progression-free and Overall Survival
Description: Probability of progression-free and overall survival after transplantation of hematopoietic cells mobilized with plerixafor
Time Frame: Day 180, 365
Population: Donor population did not receive a transplantation and therefore was not analyzed for this outcome
Measure: Number (95% Confidence Interval); unit: Percentage probability of outcome
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
Percentage probability of outcome
  Progression free survival (180 days) | 63 [46 to 79] | 69 [52 to 83]
  Progression free survival (365 days) | 53 [36 to 71] | 64 [47 to 79]
  Overall survival (180 days) | 87 [72 to 96] | 79 [63 to 91]
  Overall survival (365 days) | 63 [46 to 79] | 70 [53 to 84]
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; The probability of progression free survival and overall survival were examined in the RIC and MAC cohorts but were not directly compared between the two groups using a statistical test; Test type: Other; Kaplan-Meier curves were used to estimate the probability of progression-free survival and overall survival. Progression-free survival at 1 year was 53% (95% CI, 36% to 71%) after MAC and 64% (95% CI, 47% to 79%) after RIC. Overall survival at 1 year was 63% (95% CI, 46% to 79%) after MAC and 70% (95% CI, 53% to 84%) after RIC

12. Secondary Outcome: Cellular Composition of Allografts
Description: Cellular composition of allografts mobilized with plerixafor (stem/progenitor cells, T/B/ (Natural killer) NK-cells)
Time Frame: donation
Measure: Median (Full Range); unit: cells*10^8/kg
Arm/Group | Related Donors Receiving Plerixafor
Number analyzed (Participants) | 64
cells*10^8/kg
  CD3+ | 5.96 [2.72 to 13.0]
  CD3+CD4+ | 3.57 [2.0 to 9.4]
  CD3+CD8+ | 2.18 [0.48 to 5.0]
  CD19+ | 1.47 [0.23 to 7.43]
  CD56+ | 0.38 [0.0 to 1.10]
Statistical Analysis 1: Comparison: Related Donors Receiving Plerixafor; This outcome measure is descriptive; Test type: Other; This outcome measure is descriptive. The median cell dose and range are reported

13. Secondary Outcome: Incidence of Chronic Graft-versus-host Disease (GVHD)
Description: Incidence of chronic graft-versus-host disease (GVHD) in recipients after transplantation of hematopoietic cells mobilized with plerixafor
Time Frame: Day 365
Population: Donor arm did not receive a transplant. This group was not analyzed for graft-versus-host disease.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
Percentage of participants | 52 [33 to 70] | 39 [23 to 57]
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; The cumulative incidence of chronic graft-vs-host disease was examined in the RIC and MAC groups but was not directly compared with a statistical test; Test type: Other; The incidence of chronic GVHD was quantified by computing the cumulative incidence probability and an appropriate 95% confidence interval. Death was treated as a competing event

14. Secondary Outcome: Secondary Graft Failure After Transplantation of Hematopoietic Cells Mobilized With Plerixafor
Description: Incidence of secondary graft failure in recipients after transplantation of hematopoietic cells mobilized with plerixafor. This outcome measure is descriptive.
Time Frame: Day 365
Population: Donor population did not receive a transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients, Myeloablative Conditioning Regimen | Recipients, Reduced Intensity Conditioning Regimen
Number analyzed (Participants) | 30 | 33
Participants | 0 | 0
Statistical Analysis 1: Comparison: Recipients, Myeloablative Conditioning Regimen vs Recipients, Reduced Intensity Conditioning Regimen; Test type: Other; This is a descriptive analysis. There were no cases of secondary graft failure

15. Secondary Outcome: CD34+ Cell Count of Allografts
Description: CD34+ cell count of allografts mobilized with plerixafor
Time Frame: donation
Measure: Median (Full Range); unit: cells*10^6/kg
Arm/Group | Related Donors Receiving Plerixafor
Number analyzed (Participants) | 64
cells*10^6/kg | 4.68 [0.9 to 9.6]
Statistical Analysis 1: Comparison: Related Donors Receiving Plerixafor; Test type: Other; This outcome measure is descriptive. The median cell dose and range are reported

ADVERSE EVENTS:
Description: Recipients were not followed for adverse events.
Arm/Group | Related Donors Receiving Plerixafor
Serious Adverse Events (participants affected / at risk) | 1/64
Other Adverse Events (participants affected / at risk) | 44/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Related Donors Receiving Plerixafor (N=64)
Vasovagal reaction (Vascular disorders) | 1 (1) — One donor experienced a grade 3 vasovagal event at commencement of leukapheresis, which was unrelated to plerixafor.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Related Donors Receiving Plerixafor (N=64)
Periorbital edema (General disorders) | 1
Urticaria (General disorders) | 3
Headache (General disorders) | 9
Paresthesia (General disorders) | 17
Dizziness (General disorders) | 11
Nausea (General disorders) | 10
Vomiting (General disorders) | 3
Bloating (General disorders) | 15
Diarrhea (General disorders) | 15
Flatulence (General disorders) | 19
Abdominal pain (General disorders) | 13
Arthalgia (General disorders) | 1
Injection site reaction (Surgical and medical procedures) | 12

LIMITATIONS AND CAVEATS:
Although this was a prospective multicenter trial, conclusions are limited by the single arm design and small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No